CLINICAL TRIAL: NCT01251536
Title: A Two Arm Phase II Study of FOLFIRI in Combination With Standard or Escalating Dose of Cetuximab as First Line Treatment of K-Ras Wild Type Metastatic Colorectal Cancer: Everest 2
Brief Title: Cetuximab Standard or Dose Escalation in First Line Colorectal Cancer
Acronym: Everest2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S51532; 2009-009992-36 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; K-Ras wildtype; first line metastatic; standard cetuximab + FOLFIRI; dose escalation cetuximab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B - standard dose of cetuximab (Other): Patients with skin toxicity grade 1-4 or other significant toxicity who are not eligible for dose escalation will continue on the standard dose of cetuximab 250 mg/m2 weekly. No comparison between arms was planned.
  Interventions: Drug: Standard first line treatment with cetuximab + Folfiri
- Arm A - dose escalation of cetuximab (Experimental): Patients with skin toxicity grade 0 will follow an increasing dose schedule: on days 22 and 29 they will receive 350 mg/m2 and from day 36 onwards, 500 mg/m2 weekly.
  Interventions: Drug: Dose escalation of cetuximab

INTERVENTIONS:
Drug: Dose escalation of cetuximab — Dose, frequency & treatment mode: 400 mg/m2 (loading at day 1) followed by 250 mg/m2 weekly (at day 8 and 15)
  Arm allocation at day 22:
  Patients with skin toxicity grade 0 will follow an increasing dose schedule: on days 22 and 29 they will receive 350 mg/m2 and from day 36 onwards, 500 mg/m2 weekly
  Other Names: Erbitux
  Arms: Arm A - dose escalation of cetuximab
Drug: Standard first line treatment with cetuximab + Folfiri — Dose, frequency & treatment mode: 400 mg/m2 (loading at day 1) followed by 250 mg/m2 weekly (at day 8 and 15)
  Arm allocation at day 22:
  Patients with skin toxicity grade 1-4 or other significant toxicity who are not eligible for dose escalation will continue on the standard dose of cetuximab: 250 mg/m2 weekly.
  Other Names: Erbitux
  Arms: Arm B - standard dose of cetuximab

SUMMARY:
The purposes of this study are to determine whether administering escalating doses of cetuximab in patients with no early skin toxicity could delay the progression of disease in a significant proportion of patients and to study the molecular signatures of response.

DETAILED DESCRIPTION:
Colorectal carcinoma (CRC) is the third most common form of cancer worldwide and remains a leading malignancy both in incidence and mortality.

In the light of existing knowledge, the investigators propose a phase II open label, two arm study in patients presenting with K-Ras wild-type metastatic colorectal tumours in the first line setting. The standard combination of irinotecan plus infusional 5-FU/LV (FOLFIRI) and cetuximab will be given to all patients entering the study. As the investigators hypothesize that increasing the dose of cetuximab might increase the intensity of skin reactions that directly correlates with outcome, in patients experiencing no skin toxicity, the dose of cetuximab will be escalated from 250 mg/m2 to 350 mg/m2 and then up to 500 mg/m2, in order to better define the effect of dose escalation in the first-line setting in a K-Ras wild type tumour population and in an attempt to increase efficacy.

Pharmacokinetic studies will be performed to document PK parameters of cetuximab in patients from both arms in selected centers.

Translational research studies are planned for all patients. Some more in depth molecular testing will be performed in a subset of patients from whom three serial tissue samples from accessible metastases by biopsy are available.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (+ optional for PK and TR) must be given according to ICH/GCP and national/local regulations.
2. Patient is at least 18 years of age.
3. Patient's body weight is ≤ 120 kg.
4. Histologically proven and measurable (RECIST criteria v.1.1) metastatic adenocarcinoma of the colon or rectum, not in a previously irradiated area.
5. K-Ras wild type tumour eligible for treatment with cetuximab.
6. Unresectable metastatic disease.
7. Life expectancy of at least 12 weeks.
8. WHO ECOG performance status: 0 or 1.
9. Effective contraception for both male and female patients if the risk of conception exists.
10. Adequate organ function.
11. Adequate bone marrow, hepatic and renal function (assessed within 14 days prior to study entry):

    * Hemoglobin > 10.0 g/dL, absolute neutrophil count > 1.5 x 109/L, platelet count > 100 x 109/L
    * ALAT, ASAT < 2.5 x ULN, up to < 5 x ULN in case of liver metastases
    * Alkaline phosphatase < 2.5 x ULN
    * Total bilirubin < 1.5 x ULN
    * Creatinine clearance > 50 mL/min (calculated according to Cockroft and Gault)

Exclusion Criteria:

1. Prior treatment for metastatic disease (adjuvant therapy with fluoropyrimidines +/-oxaliplatin based regimens allowed if stopped 6 months prior to registration on study).
2. Prior treatment with EGFR inhibitor or chemotherapy with irinotecan in adjuvant settings.
3. Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to study entry.
4. Administration of any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment.
5. Concurrent chronic systemic immune therapy, chemotherapy, radiation therapy or hormone therapy not indicated in the study protocol.
6. Any active dermatological condition > grade 1.
7. Brain metastasis (known or suspected).
8. Significant impairment of intestinal absorption (e.g. chronic diarrhea, inflammatory bowel disease).
9. Other uncontrolled concomitant illness, including serious uncontrolled intercurrent infection.
10. Uncontrolled coronary artery disease and/or unstable angina, a history of a myocardial infarction within the last 12 months or heart failure NYHA class III or IV. High risk of uncontrolled arrhythmia.
11. Known allergy or any other adverse reaction to any of the drugs or to any related compound.
12. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
13. Gilbert disease.
14. Previous (within 5 years) or concurrent malignancies at other sites with the exception of surgically cured or adequately treated carcinoma in-situ of the cervix and basal cell carcinoma of the skin.
15. Organ allografts requiring immunosuppressive therapy.
16. Pregnancy (absence confirmed by serum/urine beta human choriongonadotrophin in pre-menopausal women) or breast-feeding.
17. Medical, social or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, MD, Principal Investigator — UZ Leuven
Locations (30):
- Austria (6):
  - Universitätsklinik für Innere medizin, Klinishe abteilung für hämatologie und Onkologie, Innsbruck
  - LKH Leoben, abteilung f. innere Medizin, Leoben
  - AKH Linz, Innere Medizin 3, Zentrum für Hämatologie und medizinishe Onkologie, Linz
  - Landeskrankenhaus Salzburg, Univ. Klinik für innere Medizin III, Universitätsklinikum der PMU, Salzburg
  - Krankenanstalt Rudolfstiftung, 1 medizinishe Abteilung, Vienna
  - St Vincent Krankenhaus Betriebs GmbH, Zams
- Belgium (12):
  - Imelda Ziekenhuis, Bonheiden
  - Erasme Hospital, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - AZ Middelares Gent, Ghent
  - UZ Gent, Ghent
  - Centre Hospitalier de Jolimont-Lobbes, Oncology Médicale, Haine-Saint-Paul
  - AZ Groeninge, Kortrijk
  - UZ Gasthuisberg, Leuven
  - CHC Saint Joseph, Liège
  - AZ Sint Maarten Mechelen/Duffel, Mechelen
  - H. Hartziekenhuis, Roeselare
  - AZ Turnhout (Campus St Elisabeth), Turnhout
- France (5):
  - Hôpital Avicennes, Bobigny
  - Hôpital Saint-André, Bordeaux
  - Hopital Européen Georges Pompidou, Paris
  - Centre Eugène Marquis, Rennes
  - CHU Charles Nicolle, Rouen
- Hungary (2):
  - State Health Center, Budapest
  - Medical Center of the University of Pecs , National Institute Oncology, Budapest
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clinico Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Dose Escalation of Cetuximab: Patients with no cetuximab-related skin toxicity or other significant toxicity after first 3 weeks of treatment with cetuximab standard dosing in combination with FOLFIRI, in whom cetuximab doses were increased at day 22.
  Dose escalation of cetuximab: Dose, frequency & treatment mode: 400 mg/m2 (loading at day 1) followed by 250 mg/m2 weekly (at day 8 and 15)
  Arm allocation at day 22:
  Patients with skin toxicity grade 0 will follow an increasing dose schedule: on days 22 and 29 they will receive 350 mg/m2 and from day 36 onwards, 500 mg/m2 weekly
- Arm B - Standard Dose of Cetuximab: Patients with any grade cetuximab-related skin toxicity or other significant toxicity after first 3 weeks of treatment with cetuximab standard dosing in combination with FOLFIRI, in whom cetuximab doses were maintained at standard levels at day 22.
  Standard first line treatment with cetuximab + Folfiri: Dose, frequency & treatment mode: 400 mg/m2 (loading at day 1) followed by 250 mg/m2 weekly (at day 8 and 15)
  Arm allocation at day 22:
  Patients with skin toxicity grade 1-4 or other significant toxicity who are not eligible for dose escalation will continue on the standard dose of cetuximab: 250 mg/m2 weekly.
- Not Allocated: Patients unable to continue treatment with cetuximab and FOLFIRI at standard or reduced doses, requiring discontinuation before arm allocation at day 22.
Period: Overall Study
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated
Started | 8 | 93 | 7
Completed | 8 | 93 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | Total
Number analyzed (Participants) | 8 | 93 | 7 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 69 | 5 | 76
  >=65 years | 6 | 24 | 2 | 32
Age, Continuous [Median (Full Range); unit: years] — Age at first administration of cetuximab was considered. No split per age group was performed.
  years | 66 [57 to 76] | 60 [30 to 79] | 64 [58 to 77] | 60 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 24 | 1 | 30
  Male | 3 | 69 | 6 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 4 | 0 | 4
  Belgium | 6 | 18 | 0 | 24
  Hungary | 0 | 20 | 2 | 22
  France | 0 | 5 | 2 | 7
  Spain | 2 | 46 | 3 | 51
Primary tumour [Count of Participants; unit: Participants] — Right colon= caecum, ascending and transversum colon; left colon= descending and sigmoid colon.
  Participants
    Colon right | 2 | 16 | 0 | 18
    Colon left | 2 | 47 | 5 | 54
    Rectum | 4 | 30 | 2 | 36
Tumour stage [Count of Participants; unit: Participants] — The TNM Classification of Malignant Tumors (TNM) classification is standard for describing the anatomical extent of cancers.
  "T" describes the size of the original (primary) tumor and invasion into nearby tissues. "N" describes nearby (regional) lymph nodes that are involved. "M" describes distant metastasis (spread of cancer from one part of the body to another).
  Tx: tumor cannot be assessed Tis: carcinoma in situ T0: no evidence of tumor T1, T2, T3, T4: size and/or extension of the primary tumor, where T4 is worst.
  Participants
    T1 | 0 | 2 | 0 | 2
    T2 | 0 | 2 | 0 | 2
    T3 | 2 | 46 | 2 | 50
    T4 | 4 | 27 | 4 | 35
    Tx | 2 | 16 | 1 | 19
Nodal stage [Count of Participants; unit: Participants] — TNM Classification of Malignant Tumors (TNM) classification is standard for describing the anatomical extent of cancers.
  "T" describes the size of the original (primary) tumor and invasion into nearby tissues. "N" describes nearby (regional) lymph nodes that are involved. "M" describes distant metastasis (spread of cancer from one part of the body to another).
  Nx: lymph nodes cannot be assessed; N0: no lymph nodes metastasis detected; N1: metastasis present in 1 to 3 regional lymph nodes; N2: metastasis present in more than 3 regional lymph nodes.
  Participants
    N0 | 2 | 7 | 2 | 11
    N1 | 0 | 24 | 0 | 24
    N2 | 3 | 34 | 2 | 39
    Nx | 3 | 28 | 3 | 34
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) scale measures how the disease impacts patient's daily living:
  0 Fully active, able to carry on all pre-disease performance; 1 Restricted in physically strenuous activity but able to carry out light work, e.g., house or office work; 2 Ambulatory and capable of all selfcare but unable to carry out any work; up and about more than 50% of waking hours; 3 Capable of limited selfcare; confined to bed or chair more than 50% of waking hours 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair, 5 Death
  Participants
    PS = 0 | 6 | 48 | 1 | 55
    PS = 1 | 2 | 45 | 6 | 53
Metastases [Count of Participants; unit: Participants]
  Liver only | 4 | 39 | 2 | 45
  Liver + other | 4 | 45 | 2 | 51
  Other (no liver) | 0 | 9 | 3 | 12
Index lesions [Count of Participants; unit: Participants]
  1 location | 4 | 44 | 4 | 52
  2 locations | 2 | 28 | 1 | 31
  >= 3 locations | 2 | 21 | 2 | 25
Prior cancer treatment [Count of Participants; unit: Participants]
  Chemotherapy only | 0 | 4 | 1 | 5
  Radiotherapy only | 0 | 1 | 0 | 1
  Surgery for primary tumor | 1 | 10 | 0 | 11
  Other / Combinations | 2 | 5 | 0 | 7
  No prior cancer treatment | 5 | 73 | 6 | 84
Heart rate [Mean (Full Range); unit: Bpm] | 76.7 [58 to 103] | 77.7 [44 to 105] | 84.5 [64 to 105] | 78 [44 to 105]
Systollic blood pressure [Mean (Full Range); unit: mmHg] | 120.9 [78 to 145] | 129.7 [90 to 194] | 126.6 [88 to 180] | 128.9 [78 to 194]
Diastolic blood pressure [Mean (Full Range); unit: mmHg] | 68.9 [55 to 79] | 78.8 [57 to 107] | 78.7 [61 to 105] | 78.1 [55 to 107]

OUTCOME MEASURES:

1. Primary Outcome: PFS Probability Rate at 9 Months in the Dose Escalation Arm
Description: A precise estimate (+/- 10%) of the probability of not having progression at 9 months. This measure is an estimation derived from the Kaplan-Meier algorithm and does not represent a dimple percentage of participants.
Time Frame: 9 months
Measure: Number; unit: percent probability
Groups:
- ITT / Safety Set: All patients for whom there was evidence they were administered any dose of cetuximab or FOLFIRI on study. For this study, the safety set includes all patients and is identical to the intention-to-treat (ITT) set.
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
percent probability | 45 | 48 | 0 | 55

2. Secondary Outcome: Progression Free Survival (PFS) Median Time
Description: Progression free survival time was considered from start of treatment until the first observation of disease progression or death from any cause, whichever occurred first. All patients (ITT).
Time Frame: Treatment + follow-up (3 years from database lock)
Population: All patients for whom there was evidence they were administered any dose of cetuximab or FOLFIRI on study. For this study, the safety set includes all patients and is identical to the intention-to-treat (ITT) set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
Months | 8.8 [6.2 to 25.6] | 11.5 [8.2 to 14] | 1.3 [0.9 to 1.5] | 10.7 [8.1 to 13.7]

3. Secondary Outcome: Progression Free Survival (PFS) Median Time for Resected Patients
Description: Progression free survival time was considered from start of treatment until the first observation of disease progression or death from any cause, whichever occurred first. This is the subset of resected patients (resection of secondary lesions with curative intent was performed). Patients resected after they started subsequent anti-cancer treatment or after progression on treatment were not considered as 'resected for metastatic lesions on study'. Patients were not censored at time of surgery.
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | ITT / Safety Set
Number analyzed (Participants) | 1 | 16 | 17
Months | 11.3 [0 to NA] — The upper limit of the 95%CI of the median was not determinable for Arm A. | 14.5 [12.7 to 17.9] | 14.2 [11.3 to 17.9]

4. Secondary Outcome: Progression Free Survival (PFS) Time for Resected Versus Non-resected Patients (Hazard Ratio)
Description: as for outcome 3
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
Hazard ratio | 1.17 [0.13 to 10.6] | 0.82 [0.48 to 1.42] | NA [NA to NA] — The hazard ratio and the 95%CI were not determinable for the "Not allocated" patient group. | 0.79 [0.47 to 1.34]

5. Secondary Outcome: Death Rates by 3 Years Follow-up
Description: Deaths by 3 years follow-up after last cetuximab administration + 30 days. All patients (ITT).
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
Participants
  Deceased | 6 | 65 | 7 | 78
  Alive after 3 years follow-up | 2 | 16 | 0 | 18
  Lost to follow-up before 3 years followup | 0 | 12 | 0 | 12

6. Secondary Outcome: Overall Survival (OS) Median Time
Description: Overall survival was considered from start of treatment to death. All patients (ITT).
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
months | 28.4 [12 to NA] — The upper limit of the 95%CI of the median was not determinable for Arm A. | 31.4 [25.5 to 34.9] | 4.9 [1.0 to 12.5] | 29.8 [22.4 to 33.3]

7. Secondary Outcome: Overall Survival (OS) Median Time for Resected Patients
Description: Overall survival was considered from start of treatment to death. Subset of resected patients (resection of secondary lesions with curative intent was performed). Patients resected after they started subsequent anti-cancer treatment (600-01-006 and 600-04-006) or after progression (100-02-002,
  End point description:
  Clinical trial results 2009-009992-36 version 1 EU-CTR publication date: Page 15 of 38 200-03-001, and 600-01-038) were not considered as 'resected for metastatic lesions on study.
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | ITT / Safety Set
Number analyzed (Participants) | 1 | 16 | 17
Months | NA [NA to NA] — The median and the 95%CI of the median were not determinable for Arm A. | NA [32.7 to NA] — The median and the 95%CI of the median were not determinable for Arm B. | NA [32.7 to NA] — The median and the 95%CI of the median were not determinable for the ITT set.

8. Secondary Outcome: Overall Response
Description: Overall response is defined as the best tumor response on treatment of either complete response (CR) or partial response (PR) (CR + PR). Tumor response is based on the CT/MRI assessments of target and non-target lesions as well as considering the occurrence of new lesions as per RECIST criteria. All patients (ITT).
Time Frame: Treatment duration (interval from first infusion to last infusion on study for each patient), an average of 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
Participants
  CR or PR | 6 | 64 | 0 | 70
  Other (SD, PD, not evaluable, missing) | 2 | 29 | 7 | 38

9. Secondary Outcome: Overall Response in Patients With Liver-limited Disease
Description: Overall response is defined as the best tumor response on treatment of either complete response (CR) or partial response (PR) (CR + PR). Tumor response is based on the imaging (CT/MRI) assessments of target and non-target lesions as well as considering the occurrence of new lesions as per RECIST criteria. Subset of patients with liver-limited disease.
Time Frame: Treatment duration (interval from first infusion to last infusion on study for each patient), an average of 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 4 | 39 | 2 | 45
Participants
  CR or PR | 2 | 30 | 0 | 32
  Other (SD, PD, missing) | 2 | 9 | 2 | 13

10. Secondary Outcome: Disease Control
Description: Disease control is defined as a best response on treatment (e.g. till end of treatment evaluation) of either complete response (CR), partial response (PR), or stable disease (SD) (CR + PR + SD). RECIST criteria (CT/MRI). All patients (ITT).
Time Frame: Treatment duration (interval from first infusion to last infusion on study for each patient), an average of 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
Participants
  CR, PR, or SD | 8 | 84 | 0 | 92
  Other (PD, not evaluable, missing) | 0 | 9 | 7 | 16

11. Secondary Outcome: Disease Control in Patients With Liver-limited Disease
Description: Disease control is defined as a best response on treatment (e.g. till end of treatment evaluation) of either complete response (CR), partial response (PR), or stable disease (SD) (CR + PR + SD). RECIST criteria (CT/MRI). Subset of patients with liver-limited disease.
Time Frame: Treatment duration (interval from first infusion to last infusion on study for each patient), an average of 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 4 | 39 | 2 | 45
Participants
  CR, PR, or SD | 4 | 37 | 0 | 41
  Other (PD, missing) | 0 | 2 | 2 | 4

12. Secondary Outcome: Duration of Response
Description: The duration of response in responding patients is defined as the time interval from the time measurement criteria are first met for CR/PR during treatment to either the first time disease progression is documented or death. Subset of responders.
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | ITT / Safety Set
Number analyzed (Participants) | 6 | 64 | 70
Months | 8.3 [3.6 to 24.2] | 11.7 [9.7 to 14.6] | 11.7 [8.6 to 15.4]

13. Secondary Outcome: Duration of Response in Liver-limited Disease Patients
Description: The duration of response in responding patients is defined as the time interval from the time measurement criteria are first met for CR/PR during treatment to either the first time disease progression is documented or death. Subset of responders among patients with liver-limited disease.
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | ITT / Safety Set
Number analyzed (Participants) | 2 | 30 | 32
Months | 13.9 [3.6 to 24.2] | 11.1 [7.6 to 13.0] | 11.1 [7.6 to 22.5]

14. Secondary Outcome: Resections for Metastatic Lesions
Description: All patients were deemed non-resectable at baseline but some became resectable during or posttreatment.
  All patients (ITT). Only those patients in whom resection of secondary lesions with curative intent was performed were considered as 'resected'. Patients resected after they started subsequent anti-cancer treatment (600-01-006 and 600-04-006) or after progression (100-02-002, 200-03-001, and 600-01-038) were not considered as 'resected for metastatic lesions on study'.
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
Participants
  Resected (surgery with curative intent performed) | 1 | 16 | 0 | 17
  Non-resected | 7 | 77 | 7 | 91

15. Secondary Outcome: R0 Rate (Free of Tumor After Resection for Metastatic Lesions)
Description: Rate of patients free of tumor after surgery. Subset of resected patients (resection of secondary lesions with curative intent was performed). Patients resected after they started subsequent anti-cancer treatment (600-01-006 and 600-04-006) or after progression (100-02-002, 200-03-001, and 600-01- 038) were not considered as 'resected for metastatic lesions on study'.
Time Frame: Treatment + follow-up (3 years from database lock)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | ITT / Safety Set
Number analyzed (Participants) | 1 | 16 | 17
Participants
  Free of tumor | 1 | 12 | 13
  Not free of tumor | 0 | 4 | 4

16. Secondary Outcome: Skin Toxicity (Safety)
Description: Treatment-emergent adverse events identified by the investigator as skin reaction or events with description skin infection or nail infection. Grading of severity was per NCI CTCAE version 4.0. All events are summarized based on the timing of occurrence per Arm in the first two rows, and worst grade per patient events are presented (following 3 rows). Grade 0 is the absence of any skin reaction and grade 3 is worst severity. All patients treated (Safety set).
  Note: There were 3 deviations from arm allocation rules based on the occurrence of skin toxicity. Detailed data is available upon request.
Time Frame: From signature of informed consent to last cetuximab administration on study plus 30 days for each patient, an average of 9.5 months.
Measure: Number; unit: participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated
Number analyzed (Participants) | 8 | 93 | 7
participants
  Any (onset prior to arm allocation) | 2 | 92 | 3
  Any (all times) | 7 | 93 | 3
  Grade 1 | 0 | 19 | 2
  Grade 2 | 5 | 44 | 1
  Grade 3 | 2 | 30 | 0

17. Secondary Outcome: Laboratory Safety Assessments
Description: Severe laboratory abnormalities (hematology and biochemistry grade 3 and higher). Worst grade per patient. All patients treated (Safety set).
Time Frame: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated
Number analyzed (Participants) | 8 | 93 | 7
participants
  Hemoglobin decreased | 0 | 3 | 0
  White blood cell count decreased | 3 | 8 | 0
  Neutrophils decreased | 3 | 19 | 0
  Lymphocytes decreased | 2 | 6 | 0
  Platelet count decreased | 0 | 2 | 0
  Bilirubin increased | 0 | 3 | 0
  ALAT increased | 0 | 2 | 0
  ASAT increased | 0 | 1 | 0
  ALP increased | 2 | 4 | 0
  Sodium decreased | 1 | 3 | 1
  Potassium decreased | 2 | 7 | 0
  Magnesium decreased | 1 | 2 | 0
  Magnesium increased | 0 | 1 | 0
  Serum calcium decreased | 0 | 2 | 0

18. Secondary Outcome: Deaths Till 30 Days From Last Cetuximab Administration
Description: Deaths of all causes occuring between the signature of consent and the date of last cetuximab administration + 30 days are listed per arm. None of these fatalities were deemed related to the investigational drug.
Time Frame: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated | ITT / Safety Set
Number analyzed (Participants) | 8 | 93 | 7 | 108
participants
  All causes | 1 | 6 | 2 | 9
  Colonic perforation | 1 | 0 | 0 | 1
  Malaise | 0 | 1 | 0 | 1
  Bronchial infection | 0 | 1 | 0 | 1
  Lung infection | 0 | 1 | 0 | 1
  Circulatory failure | 0 | 1 | 0 | 1
  Cardiac arrest | 0 | 1 | 0 | 1
  Colonic obstruction | 0 | 1 | 0 | 1
  Peritoneal infection | 0 | 0 | 1 | 1
  Ileus | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: From signature of informed consent to last cetuximab administration on study plus 30 days for each patient, an average of 9.5 months.
Description: SAEs occurring between the signature of the informed consent and last drug administration plus 30 days are listed. Fatalities are entered if occurred within 30 days from last drug administration. All severe AEs (grade 3-5) including SAEs, are listed in the non-serious AE table. Skin toxicity and severe lab abnormalities are further detailed in section End points.
Arm/Group | Arm A - Dose Escalation of Cetuximab | Arm B - Standard Dose of Cetuximab | Not Allocated
All-Cause Mortality (participants affected / at risk) | 1/8 | 6/93 | 2/7
Serious Adverse Events (participants affected / at risk) | 6/8 | 39/93 | 6/7
Other Adverse Events (participants affected / at risk) | 6/8 | 66/93 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Dose Escalation of Cetuximab (N=8) | Arm B - Standard Dose of Cetuximab (N=93) | Not Allocated (N=7)
Circulatory failure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 8 (8) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory insufficience (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (1)
Galbladder obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic hematoma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes angiopathy (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Severe undernutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Catheder related infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Yersinia enterocolitica gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Dose Escalation of Cetuximab (N=8) | Arm B - Standard Dose of Cetuximab (N=93) | Not Allocated (N=7)
Circulatory failure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromoembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
General deterioration (General disorders) | 0 (0) | 3 (5) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricullar fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (5) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colonic haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 14 (20) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Hepatic hematoma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fissure/feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fissure/fingers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 17 (25) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Diabetes angiopathy (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 2 (7) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Severe undernutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute cytolysis due to viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 1 (3) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 7 (16) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Yersinia enterocolitica gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Insufficient population in escalation arm A as early skin toxicity in most patients; study not powered for formal comparison between arms. Systematic error sources: some AEs re-coded by sponsor, misclassification bias (local response assessment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes